CLINICAL TRIAL: NCT04852653
Title: A Prospective Feasibility Study Evaluating Extracellular Vesicles Obtained by Liquid Biopsy for Neoadjuvant Treatment Response Assessment in Rectal Cancer
Acronym: RECC-EV
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/21
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Liquid Biopsy
Keywords: Liquid biopsy; Rectal cancer; Extracellular vesicles; Exosome; ExoDNA
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with adenocarcinoma of rectum histologically proven
  Interventions: Procedure: Supplementary blood samples collection during the normal follow up of the patients

INTERVENTIONS:
Procedure: Supplementary blood samples collection during the normal follow up of the patients — Supplementary blood samples collection during the normal follow up of the patients

SUMMARY:
Routine clinical and radiological assessment of response of patients with rectum cancer to neoadjuvant chemoradiotherapy does not allow accurate identification of complete pathological response, and leads to frequent false positive and negative results. Molecular markers reflecting the initial and post-nCRT status of the tumor would be ideal to select patients eligible for organ preservation. This project will test the detection of tumor extracellular vesicles (EVs) in liquid biopsy as a reliable marker for the identification of poor versus good responders to nCRT.

DETAILED DESCRIPTION:
Neoadjuvant treatment (NT) followed by total mesorectum excision (TME) constitues the gold standard for locally advanced carcinoma of the low and middle rectum. When good clinical response to NT is obtain, strategies with organ preservation, including close surveillance without immediate surgery or transanal local excision, can spare patients with the highly morbid and functional cost of TME. Current assessment of good responders relies on the downstaging and/or downsizing of the tumor as evaluated by MRI imaging and clinical exam. This strategy is prone to errors in more than 1/3 cases. Better assessment of tumor response to NT would better select patients eligible for organ preservation strategies. This study will use the detection of tumor extracellular vesicles (EVs) in liquid biopsy to identify good response of rectum cancer to neoadjuvant treatment. Tumor EVs will be detected in the blood of the patients at different times of their regular management (before, during and after NT). Protein content or tumor DNA in EVs will be detected after tumor DNA sequencing in the primary biopsies. Response will be assessed according to tumor EV presence or absence in the blood. As EV quantification is possible, kinetics of their detection will help response assessment and patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of rectum histologically proven
* Location ≤ 10 cm from the anal margin

  * Stage T3T4, or T2 if low rectal cancer
  * With indication of radiochemotherapy alone or chemotherapy followed by chemoradiotherapy prior to total mesorectal surgery or transanal surgery
* No metastasis
* Operable patient
* Patient ≥ 18 years old
* Patient likely to receive radiation therapy and chemotherapy.
* No history of pelvic radiotherapy for any reason
* No history of chemotherapy unless it was more than 10 years ago
* Effective contraception for patients of childbearing age: male and non-menopausal women must agree to use two medically validated methods of contraception (one for the patient and the other for the partner) during treatment and less up to 6 months for men and 4 months for women after last treatment
* Patient information and obtaining free, informed and written consent, signed by the patient and his investigator.
* Affiliate subject or beneficiary of a social security scheme of a member country of the European Community (article L1121-11 of the Code of Public Health)

Exclusion Criteria:

* Tumor of the upper rectum (> 10 cm from the anal margin)
* Metastatic disease

  . T1 stage tumor
* History of pelvic radiotherapy and chemotherapy
* Contraindication to chemotherapy and / or radiotherapy

  . Insufficient tumoral sample on initial rectal biopsy for performing molecular analysis of tumor by NGS.
* Other concomitant cancer or history of cancer other than treated in situ cervix cancer or basal cell or squamous cell carcinoma
* Pregnant woman, likely to be pregnant or breastfeeding

  * Symptomatic cardiac and / or coronary insufficiency
  * Severe renal impairment (creatinine clearance less than 30ml / min)
  * Full or partial deficiency in dihydropyrimidine dehydrogenase (DPD) (uracilemia ≥ 16 ng / ml)
  * Peripheral neuropathy> grade 1
  * Treatment with St. John's Wort
  * Treatment with yellow fever vaccine
  * Treatment with prophylactic phenytoin
  * Treatment with sorivudine or its chemically analogues related, such as brivudine
  * Active infection or other serious underlying disease likely to prevent the patient from receiving treatment
  * Persons deprived of their liberty, or under measure of judicial protection (curatorship or guardianship) or incapable of giving their consent
  * Impossibility of submitting to the medical follow-up of the test for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adenocarcinoma of rectum histologically proven
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Positivity of the liquid biopsy | 6 months
  Presence of onco-exosomes and / or exoDNA according to the response to the neoadjuvant treatment by chemotherapy alone or followed by radiochemotherapy of rectal cancer

SECONDARY OUTCOMES:
Prediction of the response of rectal cancer to neoadjuvant treatment | 6 months
  To evaluate whether the kinetics of detection of oncoexosomes and exoDNA is a predictor of the response of rectal cancer to neoadjuvant treatment
Genetic profile of the primary tumor predictive of the response to nCRT | 6 months
  To evaluate whether the initial mutational profile of the tumor is a predictor of the response of rectal cancer to chemotherapy and radiochemotherapy neoadjuvant treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No